CLINICAL TRIAL: NCT00554333
Title: An Open-label, Multi-centre, Randomised, Comparative Study of the Immunogenicity and Safety of an Inactivated Split-Virion Influenza Vaccine Administered by Intradermal Route (Flu-ID 15μg) Versus an Inactivated Adjuvanted Influenza Vaccine Administered by Intramuscular Route in Subjects 65 Years of Age or Older
Brief Title: Comparative Study of Immunogenicity and Safety of Flu-ID Vaccine Versus Flu-IM Vaccine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FID01C
Record Dates: First submitted 2007-11-05; First posted 2007-11-06 (Estimated); Last update posted 2018-03-16 (Actual); Status verified 2018-03

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Inactivated Split-Virion Influenza Vaccine for Intradermal Route
  Interventions: Biological: Flu-ID 15μg
- 2 (Active Comparator): Inactivated adjuvanted Influenza Vaccine for Intramuscular Route
  Interventions: Biological: Inactivated adjuvanted Influenza Vaccine

INTERVENTIONS:
Biological: Flu-ID 15μg — Inactivated Split-Virion Influenza Vaccine for Intradermal Route
  Arms: 1
Biological: Inactivated adjuvanted Influenza Vaccine — Inactivated adjuvanted Influenza Vaccine for Intramuscular Route
  Arms: 2

SUMMARY:
Primary objective:

* Immunogenicity To demonstrate that the influenza vaccine administered by intradermal route at least as immunogenic as the adjuvanted influenza vaccine administered by intramuscular route at the same dosage in term of HA antibody titres

Secondary objectives

* Immunogenicity

  * To describe the immune response 21 days after vaccination with the influenza vaccine administered by ID route versus the adjuvanted influenza vaccine administered by IM route..
  * To describe the compliance of both vaccines administered with the European Medicine Agency (EMEA) Note for Guidance immunogenicity criteria, specific for elderly subjects
* Safety

  - To describe the safety profile after vaccination in each group
* Acceptability

  * To describe the pain at the injection site
  * To describe the comfort of the injection

ELIGIBILITY:
Inclusion Criteria:

* Aged 65 years or older on the day of inclusion

Exclusion Criteria:

* Febrile illness (oral temperature ≥37.5°C) on the day of inclusion
* Thrombocytopenia or bleeding disorder contraindicating intramuscular vaccination
* Unstable chronic illness
* Congenital or acquired immunodeficiency,
* Any blood or blood-derived product in the past 3 months
* Current abuse of alcohol or drug addiction
* Any vaccination in the past 4 weeks or planned in the 4 weeks following study vaccination
* Any vaccination against influenza in the past 6 months
* Subjects who previously received a vaccination against influenza by intradermal route

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 795 (Actual)
Dates: Start 2007-10; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Immunogenicity Anti-Haemagglutinin (Anti-HA) antibody titres (1/dil) for the three strains obtained on Day 21 after vaccination. | 21 days

SECONDARY OUTCOMES:
Immunogenicity The derived endpoints will be: - Anti-HA individual titre ratios [Day 21 / Day 0] | 21 days
Immunogenicity The derived endpoints will be: - Seroprotection status [anti-HA individual titre ≥40 (1/dil)] on Day 21 | 21 days
Seroconversion or significant increase status at Day 21:anti-HA individual post-vaccination titre ≥40 (1/dil) on D21 for subjects with a pre-vaccination anti-HA individual titre <10 (1/dil) on D0 | 21 days
Seroconversion or significant increase status at D21: ≥4-fold increase from pre- to post-vaccination anti-HA individual titre on D21 for subjects with a pre-vaccination anti-HA individual titre ≥10 (1/dil) | 21 days
Occurrence, time to onset, number of days of occurrence, and intensity of solicited injection site adverse reactions and systemic adverse reactions occurring from D0 to D7 after vaccination | 7 days
Occurrence of some solicited adverse reactions occurring from D0 to D3 after vaccination as defined by the EMEA Note for Guidance [CPMP/BWP/214/96] | 3 days
Occurrence, nature (MedDRA PT), time to onset, duration, intensity, and relationship to vaccination (only for systemic adverse events) of unsolicited (spontaneously reported) adverse events (injection site and systemic) occurring from D0 to visit 2 | 21 days (plus or minus 3 days)
Occurrence, nature (MedDRA PT), time to onset, duration, intensity, and relationship to vaccination (only for systemic adverse events) of serious adverse events occurring from D0 to visit 2 | 21 days (plus or minus 3 days)
Intensity of pain at the time of injection evaluated just after vaccination on D0 using a Verbal Rating Scale | 1 day (day of vaccination)
Answers to the Vaccination Comfort Questionnaire completed on D21 | 21 days

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur, a Sanofi Company
Locations (8):
- Belgium (3):
  - Antwerp
  - Massemen
  - Wilrijk
- France (5):
  - Angers
  - Cherbourg
  - Laval
  - Seysses
  - Tiercé

REFERENCES:
- [Derived] Van Damme P, Arnou R, Kafeja F, Fiquet A, Richard P, Thomas S, Meghlaoui G, Samson SI, Ledesma E. Evaluation of non-inferiority of intradermal versus adjuvanted seasonal influenza vaccine using two serological techniques: a randomised comparative study. BMC Infect Dis. 2010 May 26;10:134. doi: 10.1186/1471-2334-10-134. PMID 20504306